CLINICAL TRIAL: NCT00995501
Title: The Effects of Corticosteroids, Glucose Control, and Depth-of-Anesthesia on Perioperative Inflammation and Morbidity From Major Non-cardiac Surgery (Dexamethasone, Light Anesthesia and Tight Glucose Control (DeLiT Trial))
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per interim analysis, for futility.
Sponsor: d sessler (Other)
Responsible Party: Sponsor-Investigator, d sessler, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 07-010; NCT00433251 (obsolete NCT alias)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Inflammation; Perioperative Morbidity
Keywords: steroid administration; tight glucose control; light anesthesiReducing inflammatory response to surgical stress; a
MeSH Terms: conditions — Inflammation | interventions — dexamethasone sulfate ester; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Intensive Glucose Control, Dexamethasone, light anesthesia (Active Comparator): * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Interventions: Drug: Dexamethasone Sodium Sulfate; Drug: Insulin; Drug: anesthesia management
- Intensive Glucose Control, Dexamethasone, Deep anesthesia (Active Comparator): * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Interventions: Drug: Dexamethasone Sodium Sulfate; Drug: Insulin; Other: Anesthesia management -Placebo
- Intensive Glucose Control, placebo, Light anesthesia (Active Comparator): * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Interventions: Drug: Dexamethasone Sodium Sulfate; Drug: anesthesia management; Other: Insulin - Placebo
- Conventional Glucose Control, Dexamethasone, Light anesthesia (Active Comparator): * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Interventions: Drug: Insulin; Drug: anesthesia management; Other: Dexamethasone - placebo
- Intensive Glucose Control, Placebo, Deep anesthesia (Active Comparator): * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Interventions: Drug: Dexamethasone Sodium Sulfate; Other: Insulin - Placebo; Other: Anesthesia management -Placebo
- Conventional Glucose Control, Dexamethasone, Deep anesthesia (Active Comparator): * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Interventions: Drug: Insulin; Other: Dexamethasone - placebo; Other: Anesthesia management -Placebo
- Conventional Glucose Control, Placebo, Light anesthesia (Active Comparator): * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Interventions: Drug: anesthesia management; Other: Dexamethasone - placebo; Other: Insulin - Placebo
- Conventional Glucose Control, Placebo, Deep anesthesia (Placebo Comparator): * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Interventions: Other: Dexamethasone - placebo; Other: Insulin - Placebo; Other: Anesthesia management -Placebo

INTERVENTIONS:
Drug: Dexamethasone Sodium Sulfate — 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Arms: Intensive Glucose Control, Dexamethasone, Deep anesthesia; Intensive Glucose Control, Dexamethasone, light anesthesia; Intensive Glucose Control, Placebo, Deep anesthesia; Intensive Glucose Control, placebo, Light anesthesia
Drug: Insulin — Insulin to maintain blood glucose 80-110 mg/dl.
  Arms: Conventional Glucose Control, Dexamethasone, Deep anesthesia; Conventional Glucose Control, Dexamethasone, Light anesthesia; Intensive Glucose Control, Dexamethasone, Deep anesthesia; Intensive Glucose Control, Dexamethasone, light anesthesia
Drug: anesthesia management — Light anesthesia to maintain BIS about 55
  Arms: Conventional Glucose Control, Dexamethasone, Light anesthesia; Conventional Glucose Control, Placebo, Light anesthesia; Intensive Glucose Control, Dexamethasone, light anesthesia; Intensive Glucose Control, placebo, Light anesthesia
Other: Dexamethasone - placebo — 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Arms: Conventional Glucose Control, Dexamethasone, Deep anesthesia; Conventional Glucose Control, Dexamethasone, Light anesthesia; Conventional Glucose Control, Placebo, Deep anesthesia; Conventional Glucose Control, Placebo, Light anesthesia
Other: Insulin - Placebo — Insulin to maintain blood glucose 180-200 mg/dl.
  Arms: Conventional Glucose Control, Placebo, Deep anesthesia; Conventional Glucose Control, Placebo, Light anesthesia; Intensive Glucose Control, Placebo, Deep anesthesia; Intensive Glucose Control, placebo, Light anesthesia
Other: Anesthesia management -Placebo — Deep anesthesia to maintain BIS about 35
  Arms: Conventional Glucose Control, Dexamethasone, Deep anesthesia; Conventional Glucose Control, Placebo, Deep anesthesia; Intensive Glucose Control, Dexamethasone, Deep anesthesia; Intensive Glucose Control, Placebo, Deep anesthesia

SUMMARY:
Evidence thus suggests that steroid administration, tight glucose control, and avoidance of deep anesthesia may decrease perioperative morbidity by reducing the inflammatory response to surgery. Using a three-way factorial approach, the investigators thus propose to test the primary hypotheses that major perioperative morbidity is reduced by: 1) low-dose dexamethasone; 2) intensive perioperative glucose control; and 3) lighter anesthesia.

Secondary hypotheses include that each intervention reduces circulating concentrations of the inflammatory marker CRP, and that there is a correlation between C-reactive protein (CRP) and post-operative complications. Anesthetic sensitivity predicts major and minor complications, and delirium Other secondary hypotheses are that each intervention, reduces minor surgical complications, reduces postoperative nausea and vomiting (PONV), reduces postoperative delirium, speeds hospital discharge, improves quality of life (SF-12v2 Health Survey, Christensen's VAS fatigue score), and reduces all-cause one-year mortality.

DETAILED DESCRIPTION:
The perioperative period is characterized by an intense inflammatory response marked by elevated concentrations of inflammatory markers like C-Reactive Protein (CRP). This response has been linked to increased perioperative morbidity and mortality. Available evidence suggests that blunting the inflammatory response to surgical trauma might improve perioperative outcomes. The putative benefits from blunting the surgical stress response are likely to be greatest in high-risk patients such as those having major non-cardiac surgery. We will study three interventions potentially modulating perioperative inflammation, corticosteroids, tight glucose control and light anesthesia and their effects on major morbidity and mortality resulting from major non-cardiac surgery.

Steroids are the most powerful routinely available anti-inflammatory drugs. They decrease perioperative concentrations of inflammatory markers and improve outcomes after cardiac and abdominal surgery.

Poorly controlled blood glucose worsens the inflammatory response to surgery. Hyperglycemia impairs wound healing, increases infection risk, increases overall hospital mortality, increases the risk of perioperative renal failure, and augments transfusion requirements. Treatment of hyperglycemia has been shown to improve outcomes and decrease mortality in cardiac patients. Also in critically ill patients, it decreased inflammatory markers, overall hospital mortality by 34%, blood stream infections by 46%, and acute renal failure by 41%.

Cumulative deep hypnotic time is associated with increased one-year all-cause mortality, possibly through aggravation of the inflammatory response to surgery. In contrast, avoidance of deep anesthesia appears to reduce postoperative CRP levels, the risk of nausea and vomiting, as well as postoperative hemodynamic, respiratory and infectious complications.

Evidence thus suggests that steroid administration, tight glucose control, and avoidance of deep anesthesia may decrease perioperative morbidity by reducing the inflammatory response to surgery. Using a three-way factorial approach, we thus propose to test the primary hypotheses that major perioperative morbidity is reduced by: 1) low-dose dexamethasone; 2) intensive perioperative glucose control; and, 3) lighter anesthesia.

Secondary hypotheses include that each intervention reduces circulating concentrations of the inflammatory marker CRP, and that there is a correlation between CRP and post-operative complications. Anesthetic sensitivity predicts major and minor complications, and delirium Other secondary hypotheses are that each intervention, reduces minor surgical complications, reduces postoperative nausea and vomiting (PONV), reduces postoperative delirium, speeds hospital discharge, improves quality of life (SF-12v2 Health Survey, Christensen's VAS fatigue score), and reduces all-cause one-year mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years old.
2. Major non-cardiac surgical procedures scheduled to take ≥ two hours done under general anesthesia.
3. Written informed consent

Exclusion Criteria:

1. Recent intravenous or oral steroid therapy (within 30 days); inhaled steroids are permitted
2. Any contraindications to the proposed interventions
3. ASA Physical Status > 4
4. Non English speaking patients
5. Procedures done under regional anesthesia

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2007-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basem Abdelmalak, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Abdelmalak BB, Duncan AE, Bonilla A, Yang D, Parra-Sanchez I, Fergany A, Irefin SA, Sessler DI. The intraoperative glycemic response to intravenous insulin during noncardiac surgery: a subanalysis of the DeLiT randomized trial. J Clin Anesth. 2016 Mar;29:19-29. doi: 10.1016/j.jclinane.2015.10.005. Epub 2016 Feb 2. PMID 26897443
- [Derived] Abdelmalak BB, Bonilla A, Mascha EJ, Maheshwari A, Tang WH, You J, Ramachandran M, Kirkova Y, Clair D, Walsh RM, Kurz A, Sessler DI. Dexamethasone, light anaesthesia, and tight glucose control (DeLiT) randomized controlled trial. Br J Anaesth. 2013 Aug;111(2):209-21. doi: 10.1093/bja/aet050. Epub 2013 Mar 28. PMID 23539236
- [Derived] Abdelmalak B, Maheshwari A, Kovaci B, Mascha EJ, Cywinski JB, Kurz A, Kashyap VS, Sessler DI. Validation of the DeLiT Trial intravenous insulin infusion algorithm for intraoperative glucose control in noncardiac surgery: a randomized controlled trial. Can J Anaesth. 2011 Jul;58(7):606-616. doi: 10.1007/s12630-011-9509-3. Epub 2011 May 20. PMID 21598057

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Glucose Control, Dexamethasone, Light Anesthesia: * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Dexamethasone Sodium Sulfate: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Insulin: Insulin to maintain blood glucose 80-110 mg/dl.
  anesthesia management: Light anesthesia to maintain BIS about 55
- Intensive Glucose Control, Dexamethasone, Deep Anesthesia: * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Dexamethasone Sodium Sulfate: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Insulin: Insulin to maintain blood glucose 80-110 mg/dl.
  Anesthesia management -Placebo: Deep anesthesia to maintain BIS about 35
- Intensive Glucose Control, Placebo, Light Anesthesia: * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Dexamethasone Sodium Sulfate: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  anesthesia management: Light anesthesia to maintain BIS about 55
  Insulin - Placebo: Insulin to maintain blood glucose 180-200 mg/dl.
- Conventional Glucose Control, Dexamethasone, Light Anesthesia: * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  Insulin: Insulin to maintain blood glucose 80-110 mg/dl.
  anesthesia management: Light anesthesia to maintain BIS about 55
  Dexamethasone - placebo: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
- Intensive Glucose Control, Placebo, Deep Anesthesia: * Intensive Glucose Control The target range for blood glucose will be 80-110 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Dexamethasone Sodium Sulfate: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Insulin - Placebo: Insulin to maintain blood glucose 180-200 mg/dl.
  Anesthesia management -Placebo: Deep anesthesia to maintain BIS about 35
- Conventional Glucose Control, Dexamethasone, Deep Anesthesia: * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Dexamethasone Dexamethasone administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Insulin: Insulin to maintain blood glucose 80-110 mg/dl.
  Dexamethasone - placebo: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Anesthesia management -Placebo: Deep anesthesia to maintain BIS about 35
- Conventional Glucose Control, Placebo, Light Anesthesia: * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Light anesthesia target BIS of 55
  anesthesia management: Light anesthesia to maintain BIS about 55
  Dexamethasone - placebo: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Insulin - Placebo: Insulin to maintain blood glucose 180-200 mg/dl.
- Conventional Glucose Control, Placebo, Deep Anesthesia: * Conventional Glucose Control The target range for blood glucose will be 180-200 mg/dl
  * Placebo Placebo administered at 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning.
  * Deep anesthesia target BIS of 35
  Dexamethasone - placebo: 8 mg given 1-2 hours before surgery (incision time), 4 mg on the first postoperative morning, and 2 mg on the second postoperative morning
  Insulin - Placebo: Insulin to maintain blood glucose 180-200 mg/dl.
  Anesthesia management -Placebo: Deep anesthesia to maintain BIS about 35
Period: Overall Study
Arm/Group | Intensive Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Dexamethasone, Deep Anesthesia | Intensive Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Placebo, Deep Anesthesia | Conventional Glucose Control, Dexamethasone, Deep Anesthesia | Conventional Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Placebo, Deep Anesthesia
Started | 52 | 51 | 47 | 46 | 46 | 44 | 49 | 46
Completed | 52 | 51 | 47 | 46 | 46 | 44 | 49 | 46
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Dexamethasone, Deep Anesthesia | Intensive Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Placebo, Deep Anesthesia | Conventional Glucose Control, Dexamethasone, Deep Anesthesia | Conventional Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Placebo, Deep Anesthesia | Total
Number analyzed (Participants) | 52 | 51 | 47 | 46 | 46 | 44 | 49 | 46 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 65 (11) | 64 (11) | 64 (11) | 65 (13) | 64 (11) | 63 (12) | 65 (12) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 19 | 13 | 16 | 13 | 17 | 13 | 127
  Male | 30 | 37 | 28 | 33 | 30 | 31 | 32 | 33 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 49 | 42 | 45 | 44 | 43 | 48 | 42 | 362
  African American | 2 | 2 | 5 | 1 | 2 | 1 | 1 | 4 | 18
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28 (4) | 30 (6) | 28 (6) | 28 (8) | 28 (6) | 27 (5) | 27 (6) | 29 (6) | 28 (6)

OUTCOME MEASURES:

1. Primary Outcome: Major Perioperative Morbidity
Description: Our primary outcome was a collapsed composite endpoint (any versus none) defined as the occurrence of at least one of sixteen major complications before hospital discharge, including sepsis, severe surgical site infection, myocardial infarction, heart failure, stroke, unstable ventricular arrhythmias, pulmonary embolism, pneumonia, respiratory failure, dialysis dependent renal failure, large pleural or peritoneal effusions, major bleeding, major wound and surgical site healing complications, vascular graft thrombosis, and 30-day mortality.
Time Frame: 30 day after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Dexamethasone, Deep Anesthesia | Intensive Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Placebo, Deep Anesthesia | Conventional Glucose Control, Dexamethasone, Deep Anesthesia | Conventional Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Placebo, Deep Anesthesia
Number analyzed (Participants) | 52 | 51 | 47 | 46 | 46 | 44 | 49 | 46
Participants | 10 | 10 | 8 | 9 | 10 | 8 | 11 | 9
Statistical Analysis 1: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Compare 4 arms with intensive glucose control vs. 4 arms with conventional glucose control; Test type: Superiority; p = 0.86, Regression, Logistic; Odds Ratio (OR) = 0.96, 99.6% CI 2-sided [0.45 to 2]
Statistical Analysis 2: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Compare 4 arms with Dexamethasone vs. 4 arms with Placebo; Test type: Superiority; p = 0.87, Regression, Logistic; Odds Ratio (OR) = 0.96, 99.6% CI 2-sided [0.45 to 2]
Statistical Analysis 3: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Compare 4 arms with light anesthesia vs. 4 arms with deep anesthesia; Test type: Superiority; p = 0.90, Regression, Logistic; Odds Ratio (OR) = 1, 99.6% CI 2-sided [0.49 to 2.2]

2. Secondary Outcome: 1 Year Mortality
Description: All-cause mortality
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Dexamethasone, Deep Anesthesia | Intensive Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Placebo, Deep Anesthesia | Conventional Glucose Control, Dexamethasone, Deep Anesthesia | Conventional Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Placebo, Deep Anesthesia
Number analyzed (Participants) | 52 | 51 | 47 | 46 | 46 | 44 | 49 | 46
Participants | 1 | 7 | 9 | 7 | 7 | 7 | 5 | 2
Statistical Analysis 1: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Compare 4 arms with intensive glucose control vs. 4 arms with conventional glucose control; Test type: Superiority; p = 0.8, Regression, Logistic; Odds Ratio (OR) = 0.92, 99.6% CI 2-sided [0.37 to 2.3]
Statistical Analysis 2: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Compare 4 arms with Dexamethasone vs. 4 arms with Placebo; Test type: Superiority; p = 0.84, Regression, Logistic; Odds Ratio (OR) = 1.1, 99.6% CI 2-sided [0.43 to 2.7]
Statistical Analysis 3: Comparison: Intensive Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Dexamethasone, Deep Anesthesia vs Intensive Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Dexamethasone, Light Anesthesia vs Intensive Glucose Control, Placebo, Deep Anesthesia vs Conventional Glucose Control, Dexamethasone, Deep Anesthesia vs Conventional Glucose Control, Placebo, Light Anesthesia vs Conventional Glucose Control, Placebo, Deep Anesthesia; Test type: Superiority; p = 0.87, Regression, Logistic; Odds Ratio (OR) = 1.1, 99.6% CI 2-sided [0.42 to 2.7]

ADVERSE EVENTS:
Time Frame: 1 year for all-cause mortality 30-day for major complications
Arm/Group | Intensive Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Dexamethasone, Deep Anesthesia | Intensive Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Dexamethasone, Light Anesthesia | Intensive Glucose Control, Placebo, Deep Anesthesia | Conventional Glucose Control, Dexamethasone, Deep Anesthesia | Conventional Glucose Control, Placebo, Light Anesthesia | Conventional Glucose Control, Placebo, Deep Anesthesia
All-Cause Mortality (participants affected / at risk) | 1/52 | 7/51 | 9/47 | 7/46 | 7/46 | 7/44 | 5/49 | 2/46
Serious Adverse Events (participants affected / at risk) | 10/52 | 10/51 | 8/47 | 9/46 | 10/46 | 8/44 | 11/49 | 9/46
Other Adverse Events (participants affected / at risk) | 15/52 | 25/51 | 20/47 | 17/46 | 22/46 | 21/44 | 20/49 | 24/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Glucose Control, Dexamethasone, Light Anesthesia (N=52) | Intensive Glucose Control, Dexamethasone, Deep Anesthesia (N=51) | Intensive Glucose Control, Placebo, Light Anesthesia (N=47) | Conventional Glucose Control, Dexamethasone, Light Anesthesia (N=46) | Intensive Glucose Control, Placebo, Deep Anesthesia (N=46) | Conventional Glucose Control, Dexamethasone, Deep Anesthesia (N=44) | Conventional Glucose Control, Placebo, Light Anesthesia (N=49) | Conventional Glucose Control, Placebo, Deep Anesthesia (N=46)
30-day major surgical complications (Injury, poisoning and procedural complications) | 10 (10) | 10 (10) | 8 (8) | 9 (9) | 10 (10) | 8 (8) | 11 (11) | 9 (9) — sepsis, surgical site infection, MI, heart failure, stroke, unstable ventricular arrhythmias,PE, pneumonia, respiratory failure, renal failure, large pleural/peritoneal effusions, bleeding, healing complications, vascular graft thrombosis, mortality
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Glucose Control, Dexamethasone, Light Anesthesia (N=52) | Intensive Glucose Control, Dexamethasone, Deep Anesthesia (N=51) | Intensive Glucose Control, Placebo, Light Anesthesia (N=47) | Conventional Glucose Control, Dexamethasone, Light Anesthesia (N=46) | Intensive Glucose Control, Placebo, Deep Anesthesia (N=46) | Conventional Glucose Control, Dexamethasone, Deep Anesthesia (N=44) | Conventional Glucose Control, Placebo, Light Anesthesia (N=49) | Conventional Glucose Control, Placebo, Deep Anesthesia (N=46)
30-day minor surgical complications (Injury, poisoning and procedural complications) | 15 (15) | 25 (25) | 20 (20) | 17 (17) | 22 (22) | 21 (21) | 20 (20) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes